CLINICAL TRIAL: NCT00725803
Title: A Phase 2a, Double-Blind, Randomized, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Activity of GS-9450, a Caspase Inhibitor, in Subjects With Chronic Hepatitis C (GS-US-227-0102)
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics, and Activity of GS-9450 in Subjects With Chronic HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-227-0102
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: HCV Infection
Keywords: Hepatitis C; HCV; Fibrosis; Apoptosis; GS-9450
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Subjects randomized 3:1 (active:placebo) to receive GS-9450 10 mg/day or placebo.
  Interventions: Drug: GS-9450; Drug: GS-9450 Placebo
- Cohort 2 (Experimental): Subjects randomized 3:1 (active:placebo) to receive GS-9450 40 mg/day or placebo.
  Interventions: Drug: GS-9450; Drug: GS-9450 Placebo
- Cohort 3 (Experimental): Subjects randomized 3:1 (active:placebo) to receive GS-9450 80 mg/day or placebo.
  Interventions: Drug: GS-9450; Drug: GS-9450 Placebo
- Cohort 4 (Experimental): Subjects randomized 3:1 (active:placebo) to receive GS-9450 5 mg/day or placebo. Cohort may or may not be conducted pending blinded review of previous cohorts.
  Interventions: Drug: GS-9450; Drug: GS-9450 Placebo

INTERVENTIONS:
Drug: GS-9450 — GS-9450 capsules administered orally once daily
Drug: GS-9450 Placebo — Placebo to match GS-9450 administered orally once daily

SUMMARY:
The purpose of this study is to examine the safety, tolerability, pharmacokinetics (studies how the body processes a drug), and initial activity of GS-9450 in preventing liver damage due to scarring, or fibrosis, caused by Hepatitis C Virus (HCV) infection.

DETAILED DESCRIPTION:
Approximately 32 subjects will receive GS 9450 or placebo for 14 consecutive days. Eight subjects will receive treatment within each of four dosing cohorts; 6 randomized to receive GS 9450 and two randomized to placebo:

Cohort 1: GS 9450 10 mg or placebo given daily x 14 days Cohort 2: GS 9450 40 mg or placebo given daily x 14 days Cohort 3: GS 9450 80 mg or placebo given daily x 14 days

If further characterization of the activity profile is deemed necessary, an additional cohort at a lower dose (5 mg) may be enrolled:

Cohort 4: GS 9450 5 mg or placebo given daily x 14 days

Each cohort will be conducted sequentially. Advancement to higher dose cohorts is dependent upon satisfactory safety and tolerability profiles of the preceding cohort as determined by Sponsor review (conducted in consultation with the Lead Investigator[s]). Progression to Cohort 4 (5 mg dose strength) will not require a safety review of Cohort 3 (80 mg dose strength); screening and randomization for Cohort 4 may begin immediately after fully enrolling Cohort 3. Alternatively, if a dose-response relationship is apparent in review of the blinded activity data from the first three cohorts, the final 5 mg cohort may be omitted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18 to 65 years old, inclusive.
* Willing and able to provide written, informed consent
* Have a body mass index between 19 and 32 kg/m2, inclusive, at screening.
* Have chronic hepatitis C infection of any genotype (and subtype).
* Subjects must be previously treated with pegylated interferon (PEG) or interferon (INF) with or without ribavirin (RBV) and either did not achieve a sustained viral response (undetectable HCV RNA) six months after cessation of anti-viral therapy, or did not tolerate PEG or INF with or without RBV therapy. Subjects who have contraindications to receiving PEG or INF with or without RBV may also be eligible.
* ALT >/= 1.5 X but < 10 X the upper limit of the normal range (ULN); aspartate aminotransferase (AST) < 10 X ULN; platelets >/= 75,000/mm3; total bilirubin </= 1.5 X ULN; prothrombin time </= 1.5 X ULN; albumin >/= 3.0 g/dL; absolute neutrophil count >/= 1,000 cells/mm3; and hemoglobin >/= 10 g/dL
* Creatinine clearance >/= 70 mL/min
* A female of non-childbearing potential who is documented as either surgically sterile or post-menopausal for >/= 2 years.
* Females < 2 years post-menopausal are required to have follicle-stimulating hormone (FSH) level of >/= 40 mIU/mL. If of child-bearing potential or FSH < 40 mIU/mL, must:

  1. have negative serum pregnancy test and a negative urine pregnancy test, and
  2. agree to use an acceptable method of contraception during heterosexual intercourse during the study and for >/= 30 days or one menstrual cycle (whichever is the longer) after last dose of study drug.
* If male, agree to use an acceptable method of contraception during heterosexual intercourse during the study and for at least 3 months after the last dose of study drug.
* Subjects should be in reasonably good health as determined by the Investigator.

Exclusion Criteria:

* Pregnant or breast feeding women or women who may wish to become pregnant during the study or within 30 days of study drug administration.
* Males who have partners planning to become pregnant within 30 days of study drug administration.
* Males and females of reproductive potential who are unwilling to use effective method(s) of birth control for a minimum of 30 days after ingestion of study medication
* Coinfection with hepatitis B virus (HBV) or HIV
* Known liver disease of a non-HCV etiology
* Pancreatitis
* Autoimmune disease
* History of malignancy
* Ongoing alcohol abuse.
* Recent significant infection or symptoms of infection
* Evidence of hepatocellular carcinoma (e.g., a-fetoprotein > 50 ng/mL or as indicated by recent ultrasound)
* Decompensated liver disease OR history of clinical hepatic decompensation
* Hb < 10 g/dL
* Absolute neutrophil count (ANC) < 1,000 cells/mm3
* Therapy with potentially hepatotoxic/cholestatic drugs.
* Therapy with agents having potential hepatic anti-inflammatory or anti-fibrotic properties.
* Therapy with proton pump inhibitors or histamine-2 receptor antagonists.
* Have received therapy with systemic steroids, immunosuppressant therapies or chemotherapeutic agents within 90 days prior to Day 1 or are expected to receive such therapy during the study.
* With or a history of clinically significant illness or medical disorder that may interfere with treatment, assessment or compliance.
* Have a history of a primary gastrointestinal disorder that could interfere with the absorption of the study drug or that could interfere with normal gastrointestinal anatomy or motility.
* Received study medication while participating in another research study within 60 days prior to Day 1.
* A positive urine drug screen
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients.
* Known aspirin allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Throughout 7 weeks (2 weeks on treatment and 5 weeks post-treatment)

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of GS-9450 and metabolites | 17 days (through 72 hours after last dose)
Change from baseline in alanine aminotransferase (ALT) levels at Day 14 | Day 14
Change from baseline in noninvasive markers (including cytokeratin 18 fragments) indicative of hepatic apoptosis | Through Week 5 (2 weeks on treatment and 3 weeks post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: David Oldach, MD, Study Chair — Gilead Sciences
Locations (11):
- United States (5):
  - Anaheim, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Dallas, Texas
  - San Antonio, Texas
- Germany (5):
  - Frankfurt
  - Hamburg
  - Hanover
  - Mainz
  - Würzburg
- Amsterdam, Netherlands